CLINICAL TRIAL: NCT02106429
Title: Platelet Activity in Vascular Surgery and Cardiovascular Events
Acronym: PACE
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14-00531; R01HL114978 (NIH)
Record Dates: First submitted 2014-01-22; First posted 2014-04-08 (Estimated); Results first posted 2024-07-31 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Disease; Peripheral Artery Disease; Critical Limb Ischemia
Keywords: Vascular Surgery
MeSH Terms: conditions — Cardiovascular Diseases; Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be obtained from the patient using standard aseptic phlebotomy techniques at 3 time points throughout the study. This will be pre-operatively, at post-op day 2 and at the 30-day follow up. A questionnaire, urine specimen and endothelial function test will be performed as well.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Platelet Hyperactivity: Subjects with platelet hyperactivity undergoing non emergent lower extremity revascularization.
- No Platelet Hyperactivity: Subjects with no platelet hyperactivity undergoing non emergent lower extremity revascularization.

SUMMARY:
Pathological and clinical studies have consistently demonstrated that abnormalities in thrombosis and hemostasis play a major role in the pathogenesis of atherosclerosis and atherothrombosis. Screening for abnormalities in thrombosis and hemostasis by measuring platelet activity, thrombin generation, and markers of coagulation have been proposed to identify individuals at high-risk for cardiovascular events, however, it remains a research tool not ready for implementation in standard care.

The proposed study will add to the growing understanding of platelet activity and markers of coagulation in cardiovascular disease; examine a comprehensive battery of platelet activity markers, thrombin generation, markers of coagulation, and inflammatory biomarkers in subjects undergoing vascular surgery; and will provide important data on the mechanism of increased platelet activity using micro RNA, RNA and DNA expression profiling. The study design is prospective and the main outcome measure is platelet activity measurements associated with short-term cardiovascular events in PAD patients

DETAILED DESCRIPTION:
The main aim is to determine whether preoperative platelet activity measurements are independently associated with short-term cardiovascular events in Peripheral artery disease (PAD) patients undergoing open non-emergent lower extremity vascular surgery. We will characterize the platelet phenotype in 350 PAD patients before vascular surgery and use Cox proportional hazard models to determine the independent association of the platelet phenotype with risk of cardiovascular events in the first 30 days after surgery.

Blood collection at three different time points (before surgery, following surgery while still in the hospital, and at the subjects' first return visit to the vascular surgeon following surgery) will allow us to assess the dynamic change in platelet activity, coagulation and inflammation during the perioperative period. We believe that markers of clotting and bleeding will change during the course of surgery, and that some of these markers may be used to help predict the likelihood of developing a clotting or bleeding event following surgery. The long-term goal is to develop a clinically useful assessment of platelet activity, thrombin generation, coagulation and inflammation for risk stratification that may ultimately serve as a target for therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing non emergent lower extremity revascularization
2. Use of aspirin within 48 hours prior to surgery
3. Age > 21 years of age
4. Able and willing to provide written informed consent for the study

Exclusion Criteria:

1. Use of any therapeutic anticoagulant
2. Use of any nonsteroidal antiinflammatory drug (ibuprofen, naproxen, etc.) within 72 hours
3. Thrombocytopenia (platelet count<100) or Thrombocytosis (platelet count>500)
4. Anemia (hemoglobin<9)
5. Any known hemorrhagic diathesis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study's population will be obtained form NYU Langone Medical Center, Bellevue Hospital and the VA Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2014-03; Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Berger, MD, Principal Investigator — New York University Director of Cardiovascular Thrombosis
Locations (1):
- NYU Langone Medical Center and School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Sowa MA, Hannemann C, Pinos I, Ferreira E, Biwas B, Dai M, Corr EM, Cornwell MG, Drenkova K, Lee AH, Spruill T, Reynolds HR, Hochman JS, Ruggles KV, Campbell RA, van Solingen C, Wright MD, Moore KJ, Berger JS, Barrett TJ. Tetraspanin CD37 regulates platelet hyperreactivity and thrombosis. Cardiovasc Res. 2025 Jun 12;121(6):943-956. doi: 10.1093/cvr/cvaf051. PMID 40126944
- [Derived] Dann R, Hadi T, Montenont E, Boytard L, Alebrahim D, Feinstein J, Allen N, Simon R, Barone K, Uryu K, Guo Y, Rockman C, Ramkhelawon B, Berger JS. Platelet-Derived MRP-14 Induces Monocyte Activation in Patients With Symptomatic Peripheral Artery Disease. J Am Coll Cardiol. 2018 Jan 2;71(1):53-65. doi: 10.1016/j.jacc.2017.10.072. PMID 29301628

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Platelet Hyperactivity | No Platelet Hyperactivity
Started | 203 | 43
Completed | 203 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelet Hyperactivity | No Platelet Hyperactivity | Total
Number analyzed (Participants) | 203 | 43 | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.04 (10.4) | 69.79 (10.4) | 69.89 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 12 | 76
  Male | 139 | 31 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 11 | 46
  Not Hispanic or Latino | 168 | 32 | 200
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 42 | 10 | 52
  White | 134 | 22 | 156
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 25 | 9 | 34
Region of Enrollment [Number; unit: participants]
  United States | 203 | 43 | 246

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Which Platelet Activity Measurements Were Associated With Short-term Cardiovascular Events
Description: To determine whether preoperative platelet activity measurements are independently associated with short-term cardiovascular events in Peripheral artery disease (PAD) patients undergoing open non-emergent lower extremity vascular intervention. We will characterize the platelet phenotype in 350 PAD patients before vascular surgery and use Cox proportional hazard models to determine the independent association of the platelet phenotype with risk of cardiovascular events in the first 30 days after surgery.
Time Frame: 30-days
Measure: Number; unit: participants
Arm/Group | Platelet Hyperactivity | No Platelet Hyperactivity
Number analyzed (Participants) | 203 | 43
participants | 31 | 16

ADVERSE EVENTS:
Time Frame: 30 days post surgery
Arm/Group | Platelet Hyperactivity | No Platelet Hyperactivity
All-Cause Mortality (participants affected / at risk) | 0/203 | 1/43
Serious Adverse Events (participants affected / at risk) | 0/203 | 0/43
Other Adverse Events (participants affected / at risk) | 0/203 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT02106429/Prot_SAP_000.pdf